CLINICAL TRIAL: NCT05358314
Title: Investigating Neuronal and Peripheral Markers of Brain Heart Interaction in Healthy Participants Under Stress
Acronym: HRV_DB
Status: Completed | Type: Observational
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, Joe Simon, Principal Investigator, University of Heidelberg Medical Center
Other Study IDs: S-070/2022
Record Dates: First submitted 2022-03-28; First posted 2022-05-03 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Heart Rate; Magnetic Resonance Imaging; Stress, Physiological
Keywords: fmri; heart rate variability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to investigate which regions of the brain are relevant in the regulation of cardiac control and how the interplay between HRV and those regions change during different physiological states (stress versus relaxation). In order to achieve this, we will use functional magnetic resonance imaging (fMRI) during an experimental task consisting of deep breathing and a psychosocial stress task (Montreal Imaging Stress Task).

DETAILED DESCRIPTION:
Heart rate variability (HRV) is an important indicator of an organism's ability to adapt and regulate autonomic cardiac function. High heart rate variability is an indicator of good adaptability to physical and mental demands, while decreased HRV is associated with increased vulnerability to psychological and physical stressors. Previous studies have shown that the central autonomic network, composed of several regions of the brain such as the amygdala and prefrontal cortex, play an important role in regulating heart rate variability. However, the exact neural correlates and underlying neural mechanisms involved in autonomic cardiac control are still a subject of investigation. Furthermore, the dynamic connectivity between heart rate variability and the central autonomic network under changing physiological circumstances remains largely unexplored. This study seeks to investigate which regions of the brain are especially relevant in the regulation of cardiac control and how the interplay between HRV and those regions change during different physiological states (stress versus relaxation). In order to achieve this, we will use functional magnetic resonance imaging (fMRI) during an experimental task consisting of deep breathing and a psychosocial stress task (Montreal Imaging Stress Task). This paradigm will allow assessing the dynamic interplay between the heart and the brain. 30 healthy participants will be recruited, in addition to fMRI scanning participants will perform a psychometric test battery. A better understanding of these psychobiological mechanisms is a fundamental requirement for a better understanding of the autonomic regulation of HRV and the development of improved treatment strategies for disorders characterized by an impaired autonomic system and reduced HRV.

ELIGIBILITY:
Inclusion Criteria:

1. Over age of 18 years.
2. Right-handedness.
3. Normal or corrected-to-normal vision.

Exclusion Criteria:

1. History of head injury or surgery
2. History of neurological disorder
3. Severe psychiatric comorbidity (psychosis, bipolar disorder, substance abuse)
4. Smoking
5. Borderline personality disorder
6. Current psychotropic medication
7. Inability to undergo fMRI scan (e.g. metallic implants, claustrophobia, pacemakers)
8. Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Experimental fMRI task (Stress induction following paced breathing) | 30 minutes
  Participants are instructed to breathe at a very low pace and then have to complete an arithmethic task designed to induce stress.
HRV reactivity during stress | 30 minutes
  Heart Rate Variability is assessed during MRI scanning using plethysmography.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany